CLINICAL TRIAL: NCT06540287
Title: An Observational Study of Aging Biomarkers in Older Elite Athletes Compared to Non-exercising Healthy Older Adults.
Brief Title: Molecular Optimization Via Exercise (MOVE)
Status: Recruiting | Type: Observational
Sponsor: Buck Institute for Research on Aging (Other)
Responsible Party: Sponsor
Other Study IDs: BUCK_2401
Record Dates: First submitted 2024-07-26; First posted 2024-08-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Aging
Keywords: Biomarkers; Healthy older adults; Older elite athletes
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma Serum White Blood Cells Muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 cohort: Healthy Older Adults (HOA): This cohort will include healthy older adults, aged 65y or over, who participate in less than 60 minutes of structured exercise each week.
  Interventions: Other: Observational
- Group 2 cohort: Elite Older Athletes (EOA): This cohort will include healthy older adults, aged 65y or over, who are elite athletes for their age (determined by interview and VO2max)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention

SUMMARY:
This study is to investigate characteristics of muscle, blood, and urine samples from older adults (ages 65-80) who are either sedentary or athletes performing at an elite level for their age. This observational study will include bio-specimen collection, as well as physical and cognitive function testing and body composition.

DETAILED DESCRIPTION:
The study will enroll a total of 80 subjects-20 of each gender for each cohort. Participation in the study involves 3 visits that must take place within 12 weeks. Optional l follow up visits may be completed at 12- and 24- months after completion of the main study.

The first visit is a screening and enrollment visit. At this visit, informed consent will be obtained and a detailed medical history, screening blood sample collected, and physical assessment will be performed (including, but not limited to vital signs, resting ECG, body composition). Additionally, an exercise history interview will be performed to assess for cohort eligibility. Participants will be familiarized with testing equipment during the screening visit and will perform the Astrand-Rhyming submaximal bicycle test. A short physical function testing battery will be performed, including the short physical performance battery, 6 minute walk test, grip strength, 1 rep max leg press, and leg press fatigue testing.

The second visit will include maximal exercise testing, quality of life assessment, and cognitive function testing. Participants will be allocated into their cohort at this visit.

The third visit will include thigh muscle sample collection via needle biopsy and blood sample collection.

ELIGIBILITY:
1. Willing and able to provide consent to take part in the MOVE-1 Main Study.
2. Willing and able to attend study visits and comply with all procedures of study data collection visits.
3. Able to read and speak English well enough to provide informed consent and understand instructions.
4. Healthy adults between the age of 65 - 80 y.
5. BMI >19 to < 35 kg/m2
6. No personal plans (i.e., vacations or medical procedures) during the expected study period (Screening, Test Visit 1, 2 and Sample Collection Visit).
7. Older Elite Athletes (OEA):

   • Evidence of current physical activity at an elite level for their age, as well as a consistent history of high activity level. This is assessed by interview, review of training data and/or competition results, and by review of the VO2 max data obtained during Testing Visit 1.
8. Healthy Older Adults (HOA):

   * Sedentary, defined as self-reporting no more than 1 day per week, lasting no more than 60 minutes, of regular (structured) endurance exercise [e.g., brisk walking, jogging, running, cycling, elliptical, or swimming activity that results in feelings of increased heart rate, rapid breathing, and/or sweating] or resistance exercise (resulting in muscular fatigue) in the past year.
   * Persons bicycling as a mode of transportation to and from work >1 day/week etc. are not considered sedentary.
   * Leisure walkers are included unless they meet the heart rate, breathing, and sweating criteria noted above.
   * Does not have a physically active job, no history of physically active job (i.e., postal worker, fire officer
   * No history of consistent high activity level (meeting above criteria) in the last 25 y.

3.2.2. Main Study Exclusion Criteria

1. Subject requires assistance with any activity of daily living, excluding continence.
2. Subject lives in an institutional setting (skilled nursing facility or residential care facility for the elderly).
3. Abnormal bleeding or coagulopathy (self-report): History of a bleeding disorder, wound healing disorder or clotting abnormality.
4. Female participants must be post-menopause.
5. Musculoskeletal conditions that would prevent completion of any required exercise testing.
6. Elevated blood pressure readings (screening test): Resting Systolic Blood Pressure (SBP) ≥150 mmHg or resting Diastolic Blood Pressure (DBP) ≥90 mmHg
7. Diabetes (self-report and screening tests): Treatment with any hypoglycemic agents (self-report), fasting glucose >125 mg/dL (screening test; may reassess once), use of hypoglycemic drugs for non-diabetic reasons (self-report).
8. Pulmonary (self-report): Clinical diagnosis of any chronic pulmonary disease that limits exercise capacity.
9. Cardiovascular (self-report, screening test, and clinician judgement): Congestive heart failure, coronary artery disease, significant valvular disease, congenital heart disease, serious arrhythmia, pulmonary embolism, stroke, or symptomatic peripheral artery disease (self-report, screening test). Specific criteria used to determine whether a volunteer can undergo the screening CPET follow the American Heart Association (AHA) Criteria [6]. Inability to complete the CPET. Reassessment of the CPET may be allowed under some circumstances (e.g., test was not a maximal effort)
10. Abnormal blood lipid profile (screening test): Fasting triglycerides >500 mg/dL. Low-density lipoprotein cholesterol (LDL-C) >190 mg/dL
11. Cancer (self-report): History of cancer treatment (other than non-melanoma skin cancer, or chronic lymphocytic leukemia) and not "cancer-free "for at least 2 years. Anti-hormonal therapy (e.g., for breast or prostate cancer) within the last 6 months.
12. Chronic active or latent infection (self-report): Active or latent infections requiring chronic antibiotic or anti-viral treatment, excluding herpes simplex virus. Chronic active infection whether on chronic antimicrobials or not. Human Immunodeficiency Virus. Active hepatitis B or C undergoing antiviral therapy. Individuals successfully treated for hepatitis C and virologically negative for at least 6 months are not excluded.
13. Liver enzyme tests (alanine transaminase, aspartate transaminase) (screening test): >2 times the laboratory upper limit of normal. Reassessment during screening may be allowed under some conditions (e.g., recent use of acetaminophen). Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting.
14. Chronic renal insufficiency (screening test): Estimated glomerular filtration rate <60 mL/min/1.73 m2 from serum creatinine (mg/dL) by the Chronic Kidney Disease Epidemiology Collaboration equation. Subjects must be able to produce urine. Reassessment may be allowed under some conditions (e.g., questionable hydration status or other acute renal insult)
15. Hematocrit (screening test): Hematocrit >3 points outside of the local normal laboratory ranges for women and men. Reassessment may be allowed under certain conditions. Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting.
16. Blood donation (self-report): Whole blood donation in the last 3 months or plans for blood donation during the entire protocol period. Platelet or plasma donation in the last week or plans for platelet or plasma donation during the entire protocol period.
17. Autoimmune disorders (self-report): Individuals receiving any active systemic treatment (including immunosuppressants and/or monoclonal antibodies) within the last 6 months.
18. Alcohol consumption (self-report): Current consumption of more than 7 drinks per week for women More than 14 drinks per week for men. History of binge drinking in the past five years (≥5 drinks for males or ≥4 drinks for females in a 2-hour period more than once per month)
19. Tobacco (self-report): Current smokers: any tobacco or e-cigarette/e-nicotine products. Former smokers: Stopped smoking <10 years at time of screening for those with a ≥20 pack-year smoking history. Stopped smoking <5 years at time screening for those with a <20 pack-year smoking history.
20. Recreational drug use (self-report): Self-reported use ≥3 days/week in any form
21. Shift workers (self-report): Night shift work in the last 6 months. Planning night shift work during the study period.
22. Cognitive status (screening): Unable to give consent to participate in and safely complete the protocol, as based on the judgement of the investigators.
23. Psychiatric illness (self-report and screening test): Hospitalization for any psychiatric condition within one year (self-report).
24. Weight change (self-report): Weight change (intentional or not) over the last 2 months of >5% of body weight. Plan to lose or gain weight during the study
25. Lidocaine or other local anesthetic allergy (self-report): Known allergy to lidocaine or other local anesthetic
26. COVID-19 infection: Individuals who tested positive for COVID-19 but were not hospitalized must be symptom free, at least 14 days (without a negative antigen test) or symptom-free at least 7 days with a negative antigen test on the day of the study visit. A PCR test can be used if antigen tests are not available.
27. Other (clinician judgement): Genetic metabolic disorders that could affect metabolomic results (e.g., phenylketonuria). Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric, metabolic, or other conditions that, in the opinion of the local clinician, would preclude participation and successful completion of the protocol. Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Male and female Older Endurance Athletes (OEA) at/over the age of 65 - 80 y (exercising at an elite level for their age - assessed by interview and review of training data and competition/results)
  Male and female Healthy Older Adults (HOA) at/over the age of 65 -80 y who do not regularly exercise (no more than one day per week lasting no more than 60 mins of regular structured exercise)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Muscle cellular aging - spatial transcriptomics | Day 2
  Differences between athletes and sedentary in muscle spatial transcriptomic between OEA and HOA groups
Muscle cellular aging - single cell transcriptomics | Day 2
  Differences between athletes and sedentary in muscle single cell transcriptomic between OEA and HOA groups

SECONDARY OUTCOMES:
Differences between concentration of proteins in the muscle | Day 2
  Proteomic analysis to measure differences in protein abundance in EOA vs HOA
Differences between concentration of metabolites in the muscle | Day 2
  Metabolomic analysis to measure differences in metabolite abundance in EOA vs HOA
Differences between function of muscle mitochondria | Day 2
  Analysis of respiratory function of isolated mitochondria
Blood metabolites | Day 2
  Metabolic analysis: differences between athletes and sedentary in blood metabolites
Blood proteins | Day 2
  Proteomic analysis: differences between athletes and sedentary in blood protein concentration
Blood cell immune function | Day 2
  Differences between athletes and sedentary in blood cell immune function
Blood cell gene expression | Day 2
  Differences between athletes and sedentary in blood cell gene expression
Urine metabolites | Day 2
  Differences between athletes and sedentary in urine metabolites
Physical function - VO2 max | Day 1
  Oxygen uptake measured during a ramp test on a bicycle ergometer
Physical function - grip strength | Day 1
  Measured in both hands using a dynamometer
Physical function - 6 minute walk test | Day 1
  Measure distance covered in 6 minutes on an indoor walk track
Physical function - short physical performance battery | Day 1
  SPBB includes balance, gait speed and chair sit tests, consolidated to one score
Physical function - leg strength | Day 1
  Maximal leg press weight will be determined on a gym machine via progressive increases in weight
Physical function - leg press fatigue | Day 1
  70% of the maximal leg press weight will be used. Subjects will complete as many repetitions as possible of the 70% weight and number of repetitions will be recorded.

OTHER OUTCOMES:
Body composition - BIA | Day 1
  Body composition measured by bioelectrical impedance
Body composition - muscle mass | Day 2
  Total muscle mass measured by D3 creatine supplement followed by urine collection
Cognitive function - Montreal Cognitive Assessment | Day 1
  Paper and interview based test that measures multiple domains of function
Cognitive function - digit symbol substitution | Day 1
  Paper based test that involves matching symbols and numbers in a set time.
Cognitive function - trails A and B | Day 1
  Paper based test that involves joining numbers or numbers and letters in series, as fast as possible.
Social determinants of health | Day 1
  Assessed by Upstream Risks paper based self-complete questionnaire
Sleep quality questionnaire | Day 1
  Pittsburgh Sleep Quality Index assessed by paper based self-complete questionnaire
Overal function perception | Day 1
  SF-36 (Short Form 36) validated questionnaire (paper based, self complete) that determines ease of completion of different life activities.
Depression | Day 1
  Geriatric Depression Scale (GDS) validated questionnaire (paper based, self complete) that assesses presence of depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: John C Newman, MD PhD, Principal Investigator — Buck Institute
Locations (1):
- Buck Institute for Research on Aging, Novato, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harridge SD, Lazarus NR. Physical Activity, Aging, and Physiological Function. Physiology (Bethesda). 2017 Mar;32(2):152-161. doi: 10.1152/physiol.00029.2016. PMID 28228482
- [Background] Duggal NA, Pollock RD, Lazarus NR, Harridge S, Lord JM. Major features of immunesenescence, including reduced thymic output, are ameliorated by high levels of physical activity in adulthood. Aging Cell. 2018 Apr;17(2):e12750. doi: 10.1111/acel.12750. Epub 2018 Mar 8. PMID 29517845